CLINICAL TRIAL: NCT06375226
Title: Autism Spectrum Disorder and Attachment. An Explorative Study of Attachment Styles in Adults With Autism Spectrum Disorder
Brief Title: Autism and Attachment. An Explorative Study of Attachment Styles in Autistic Adults.
Acronym: ASDA
Status: Recruiting | Type: Observational
Sponsor: Parnassia Groep (Other)
Responsible Party: Principal Investigator, Stephanie Bohnen, Principal Investigator, Parnassia Groep
Other Study IDs: 2023.17; 2023.0871 (Other: METC Amsterdam UMC)
Record Dates: First submitted 2024-04-16; First posted 2024-04-19 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; Attachtment; Adults
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The present study examines the relationship between attachment and autism spectrum disorder (ASD) in adults.

DETAILED DESCRIPTION:
Rationale: Previous research on autism spectrum disorder (ASD) and attachment has improved understanding of the aetiology and development of the disorder. Research on adults with ASD, however is scarce. The study is focussed on attachment in adults with ASD. Objective: The aim of the current study is to explore attachment styles of adults with ASD and examining the relationship between attachment and ASD.

The study requires 60 participants.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria are:

  * a primary clinical diagnosis of DSM-5 ASD (APA, 2013)
  * age 18 - 65 years
  * no intellectual disability (IQ > 80)

Exclusion Criteria:

* acute psychosis
* acute suicidality
* psychotic disorder
* intellectual disability (IQ < 80)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults (>18 years) with ASD, and without intellectual disability. Participants will be recruited from SARR Autism Rotterdam and Antes, both part of Parnassia Group in the Netherlands. SARR Autism Rotterdam is specialized in psychodiagnostic assessments and interventions for children, adolescents, and adults with ASD. Antes and Parnassia Group are multisite mental health institutes specialized in psychodiagnostic assessments and interventions for adults with a broad range of psychiatric disorders, including ASD.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
The Social Responsiveness Scale - Adult version (SRS-A) | 15 minutes
  The SRS-A is a screening tool for identifying possible ASD characteristics in adults suspicious for ASD, is 64-item self-report questionnaire measuring various dimensions of interpersonal behavior, communication, and rigid, repetitive behaviour and interests, characteristic for adults with ASD. Each item is rated on a 1-4 point scale.
The Attachment Styles Questionnaire (ASQ) | 15 minutes
  The ASQ is a questionnaire consisting of 24 items and assesses four attachment styles (secure, preoccupied, fearful, and dismissing). The 5-point rating scale ranges from 1 (strongly disagree) to 5 (strongly agree).
Experiences in Close Relationships - Revised questionnaire (ECR-r) | 15 minutes
  The ECR-r measures adult attachment within romantic relationships in past and present in 36 items, consisting of two subscales of 18 items each (attachment anxiety and attachment avoidance). Each item is rated from 'strongly disagree' (1) to 'strongly agree' (7).

CONTACTS AND LOCATIONS:
Overall Officials: Richard Vuijk, Dr., Principal Investigator — Parnassia Groep Antes
Locations (1):
- ParnassiaGroep Antes, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-19): https://cdn.clinicaltrials.gov/large-docs/26/NCT06375226/Prot_SAP_000.pdf